CLINICAL TRIAL: NCT05139797
Title: Artificial Intelligence Guided Echocardiographic Screening of Rare Diseases
Brief Title: Artificial Intelligence Guided Echocardiographic Screening of Rare Diseases (EchoNet-Screening)
Status: Recruiting | Type: Observational
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Lily Stern, Staff Physician, Cedars-Sinai Medical Center
Other Study IDs: STUDY00001720
Record Dates: First submitted 2021-11-18; First posted 2021-12-01 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Cardiac Amyloidosis
Keywords: Echocardiogram; Artificial Intelligence
MeSH Terms: conditions — Amyloid Neuropathies, Familial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

GROUPS / COHORTS (1):
- Artificial Intelligence Screening for Cardiac Amyloidosis: An artificial intelligence algorithm will produce a probability of cardiac amyloidosis that will trigger referral to specialty clinic for further evaluation.
  Interventions: Other: EchoNet-LVH screening for cardiac amyloidosis

INTERVENTIONS:
Other: EchoNet-LVH screening for cardiac amyloidosis — An AI algorithm identifies LVH, low voltage, and high suspicion for cardiac amyloidosis. The intervention is the suspicion score. Patients with high suspicion score will be referred to specialty clinic for standard of care evaluation, screening, and treatment as determined by physicians.

SUMMARY:
Despite rapidly advancing developments in targeted therapeutics and genetic sequencing, persistent limits in the accuracy and throughput of clinical phenotyping has led to a widening gap between the potential and the actual benefits realized by precision medicine.

Recent advances in machine learning and image processing techniques have shown that machine learning models can identify features unrecognized by human experts and more precisely/accurately assess common measurements made in clinical practice.

The investigators have developed an algorithm, termed EchoNet-LVH, to identify cardiac hypertrophy and identify patients who would benefit from additional screening for cardiac amyloidosis and will prospectively evaluate its accuracy in identifying patients whom would benefit from additional screening for cardiac amyloidosis.

DETAILED DESCRIPTION:
Despite rapidly advancing developments in targeted therapeutics and genetic sequencing, persistent limits in the accuracy and throughput of clinical phenotyping has led to a widening gap between the potential and the actual benefits realized by precision medicine. This conundrum is exemplified by current approaches to assessing morphologic alterations of the heart. If reliably identified, certain cardiac diseases (e.g. cardiac amyloidosis and hypertrophic cardiomyopathy) could avoid misdiagnosis and receive efficient treatment initiation with specific targeted therapies. The ability to reliably distinguish between cardiac disease types of similar morphology but different etiology would also enhance specificity for linking genetic risk variants and determining mechanisms

Recent advances in machine learning and image processing techniques have shown that machine learning models can identify features unrecognized by human experts and more precisely/accurately assess common measurements made in clinical practice. In echocardiography, this ability for precision measurement and detection is important in both disease screening as well as diagnosis of cardiovascular disease.

Echocardiography is routinely and frequently used for diagnosis and prognostication in routine clinical care, however there is often subjectivity in interpretation and heterogeneity in application. Human attention is fatigable and has heterogenous interpretation between providers. AI guided disease screening workflows have been proposed for rare diseases such as cardiac amyloidosis and other diseases with relatively low prevalence but significant human impact with targeted therapies when detected early. This is an area particularly suitable for AI as there are multiple mimics where diseases like hypertrophic cardiomyopathy, cardiac amyloidosis, aortic stenosis, and other phenotypes might visually be similar but can be distinguished by AI algorithms. The investigators have developed an algorithm, termed EchoNet-LVH, to identify cardiac hypertrophy and identify patients who would benefit from additional screening for cardiac amyloidosis, hypertrophic cardiomyopathy and other diseases. E

ELIGIBILITY:
Inclusion Criteria:

* Patients who have a high suspicion for cardiac amyloidosis by AI algorithm

Exclusion Criteria:

* Patients who decline to be seen at specialty clinic
* Patients who have passed away

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have a high suspicion for cardiac amyloidosis by AI algorithm
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-11-18 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Number of New Diagnoses of Cardiac Amyloidosis Found | 6 months
  From chart review, identification of patients who have a downstream diagnosis of cardiac amyloidosis

SECONDARY OUTCOMES:
Number of New Diagnoses of TTR Amyloidosis Found | 6 months
  From chart review, identification of patients who have a downstream diagnosis of TTR amyloidosis
Number of New Diagnoses of AL Amyloidosis Found | 6 months
  From chart review, identification of patients who have a downstream diagnosis of AL amyloidosis

CONTACTS AND LOCATIONS:
Locations (1):
- Cedars-Sinai Medical Centre (Los Angeles), Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://arxiv.org/abs/2106.12511